CLINICAL TRIAL: NCT01326923
Title: Phase II Trial of Induction Chemotherapy (ICT) Followed by Concurrent Chemoraditherapy (CR) With Monoclonal Antibody Cetuximab in Locally Advanced Head and Nec Squamous Cell Cancer
Brief Title: Induction Chemo Then Concurrent Chemoradiotherapy With Cetuximab in Locally Advanced Head and Neck Squamous Cell Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principle Investigator left the institution.
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Glenn Mills, Director, FWCC, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-109
Record Dates: First submitted 2011-03-24; First posted 2011-03-31 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: Head; Neck; Locally advanced; Squamous Cell; Hypopharynx; Larynx; Oral Cavity; Base of Tongue; Tonsil; Neck lymph node; Resection
MeSH Terms: conditions — Laryngeal Diseases | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): Single arm Phase II Study Induction Chemo then Concurrent Chemoradiotherapy with Cetuximab in Locally Advanced Head and Neck Squamous Cell Cancer
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Single arm phase II study of chemotherapy
  Other Names: Single arm phase II study

SUMMARY:
This is an open label, single arm Phase II study of induction chemotherapy followed by concurrent chemo-radiotherapy in patients with locally advanced head and neck squamous cell cancer (HNSCC) using monoclonal antibody cetuximab. Those patients with locally advanced HNSCC deemed to be candidates for definitive concurrent chemo-radiotherapy will be treated initially with 6 weeks of PCC (Paclitaxel, cetuximab and Carboplatin). This will be followed by a week of no treatment for interim evaluation, followed by definitive concurrent chemo-radiotherapy using 70Gy radiation with weekly cetuximab and cisplatin for 7 weeks. The hypothesis of the study is that the use of cetuximab during induction chemotherapy followed by cetuximab concurrent with chemoradiotherapy using low dose weekly cisplatin will improve local control as well as distant spread.

DETAILED DESCRIPTION:
Chemotherapy:

Chemotherapy would be used in two phases. In the initial phase all patients would be treated with ICT involving 6 cycles of PCC. This involves Cetuximab 400mg/m2 Week 1 and then 250mg/m2 weekly, Paclitaxel 80mg/m2 weekly and carboplatin AUC 2 weekly for 6 weeks followed by concurrent chemoradiotherapy with cetuximab. After ICT patients would be given weekly Cisplatin at 30mg/m2 and cetuximab at 250mg/m2 concurrent with radiation therapy.

Radiation Therapy:

Typically for tumors treated by megavoltage (6MV) radiotherapy alone or with chemotherapy, the primary tumor bed with an adequate margin and the draining lymphatics will be treated with parallel opposed lateral treatment portals; the lower neck node bearing area will be treated through an anterior port. The standard total dose for the targeted tumor bed and electively treated lymphatics is 50 Gy/25 fractions, and then, an additional boost dose to the neoplasm-bearing site(s) of 16 Gy to 20 Gy.

The total dose received by the spinal cord should not be allowed to exceed 46 Gy. For N1 to N3 disease, they also shall need a total dose (boost included) of 66 Gy and perhaps up to 70 Gy if it can be safely given 6.4 Study Outline:

1. Patients who are deemed eligible and sign informed consent would be enrolled in the clinical trial.
2. Prior to starting therapy staging PET/CT scan, medical history, physical exam, hematologic and biochemical testing will be undertaken.
3. Since mucositis and oropharyngeal dysfunction is very likely with chemo-radiation PEG tube placements will be considered prior to treatment, in order to allow adequate nutrition in case of mucositis.
4. Prior to starting radiation patients would undergo dental evaluation which is a standard practice.
5. Patients would then undergo 6 weeks of ICT using PCC. Based on toxicity dose would be modified as described in section 8.
6. For PCC regimen, cetuxmiab would be given first followed by paclitaxel and then carboplatin using standard pre-medication.
7. A CT scan (no PET scan) of the head and neck will be performed during the evaluation Week 7 on any day of that week.
8. Following induction chemotherapy patients would be treated with radiation therapy of up to 70 Gy concurrent with weekly Cisplatin at 30mg/m2 and cetuximab at 250mg/m2 for the duration of radiation therapy. Again dose modifications would be performed based as described in section 8.
9. Cetuximab would be administered first followed by cisplatin concurrent with radiation.
10. History and Physical examination would be performed at the end of treatment to document response and assess toxicity

10. Patient with residual disease at the primary site or neck after completion of chemoradiotherapy would be offered surgery.

11. Week 26 (3 months) after completion of radiation therapy a repeat PET scan will be performed to assess response which is standard of care.

12. After completion of all treatment patients will be followed at every 3 months interval to document relapse or manage toxicities from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years and older with histologically proven locally advanced stage III or IV unresectable Squamous cell head and neck cancer SCCHN (including cancers of oral cavity, oropharynx, larynx and hypopharynx) with no evidence of distant metastasis
2. A careful evaluation for resection is required from the surgeon and criteria for unresectability carefully defined for individual primary sites as follows:

   * Hypopharynx: The tumor must extend across the midline of the posterior pharyngeal wall or be fixed to the cervical spine
   * Larynx: There must by either direct extension into surrounding muscle or skin or greater than 3 cm of sub-glottic extension
   * Oral cavity: The lesion must be so extensive that a functional reconstruction is not possible.
   * Base of Tongue: The tumor must extend into the roof of tongue, or the patient must refuse a recommended total glossectomy
   * Tonsil: The tumor must extend into the pterygoid region as manifested by clinical trismus or demonstrated across the midline of the pharyngeal wall or directly into soft tissue of the neck
   * Patients with neck lymph node metastases fixed to the carotid artery, the mastoid, the base of the skull, or the cervical spine are considered un-resectable
   * Medical unsuitability for resection is not sufficient for patient eligibility
   * Patient's refusal for surgery except in case of total glossectomy is not considered a reason for unresectibility
3. Patients must have received no prior treatment for head and neck cancer
4. ECOG Performance status 0-1
5. Adequate organ function (All labs should be obtained within 14 days prior to start of study drug treatment)

   * leukocytes > 3,000/mcL
   * absolute neutrophil count > 1,500/mcL
   * platelets > 100,000/mcL
   * total Bilirubin within normal institutional limits
   * AST (SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
6. Ability to give informed consent and willingness to adhere to study protocol
7. Subjects of reproductive potential must agree to follow accepted birth control methods during treatment and for 12 months after completion of treatment. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study

Exclusion Criteria:

1. Patient who have had prior treatment for head and neck cancer
2. Prior history of radiation to head and neck area
3. Known malignancy other than the current cancer
4. Uncontrolled intercurrent illness including but not limited to ongoing active infection, history of cardiac disease, e.g. uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within last six months or ventricular arrhythmias requiring medication, psychiatric illness that would impair patients ability to comply with study requirements
5. Pregnant or lactating women (any women becoming pregnant during the study will be withdrawn from the study)
6. Patient with documented or symptoms of peripheral neuropathy
7. History of allergic reaction to compounds similar to the ones used in this study
8. Any condition that would hamper ability to give informed consent or ability to comply with study protocol
9. HIV patients on anti-retroviral therapy are in-eligible to participate in this study because of potential interaction with the study drugs and increase susceptibility for infections during course of marrow suppressive chemotherapy and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syed H Jafri, MB,B,S, Principal Investigator — LSU shreveport
Locations (1):
- LSU Health Sciences Center, Shreveport, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 48 [40 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Analysis at Week 26
Population: The Principal Investigator left the institution. Despite exhausting all efforts to contact the Responsible Party and study team members to retrieve the collected data, or to have them enter the data, efforts were unsuccessful, and no data are available to be reported
Arm/Group | Single Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival
Description: Improvement in progression free survival (PFS)in locally advanced stage III and IV head and neck cancer patients with sequential (ICT) followed by Concurrent chemo-radiotherapy (CR) using monoclonal antibody Cetuximab as compared to historical controls.
Time Frame: Analysis at Week 26
Population: as for outcome 1
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=7)
shingles (Infections and infestations) | 1 (1)
hospitalizations (Gastrointestinal disorders) | 1 (2) — nausea, vomiting, diarrhea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes